CLINICAL TRIAL: NCT06033586
Title: An Extension Study to Evaluate the Long-term Safety of Rusfertide (PTG-300) in Subjects With Polycythemia Vera (THRIVE)
Brief Title: Study to Evaluate the Long-term Safety of Rusfertide (PTG-300) in Subjects With Polycythemia Vera
Acronym: THRIVE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTG-300-21
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Intervention Model Description: Open-label rusfertide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label rusfertide (Experimental): Open-label rusfertide
  Interventions: Drug: Open-label rusfertide

INTERVENTIONS:
Drug: Open-label rusfertide — subcutaneous rusfertide

SUMMARY:
The goal of this clinical trial is to assess long-term safety and efficacy of rusfertide in subjects with polycythemia vera. Subjects who complete dosing with rusfertide until the end-of-treatment visit of a Phase 2 rusfertide study and meet the inclusion/exclusion criteria for this study, are eligible to participate in this open-label study and continue treatment with rusfertide.

DETAILED DESCRIPTION:
This is an open-label study designed to assess the long-term safety and efficacy of rusfertide. This study aims to provide long-term rusfertide treatment to subjects who complete dosing until the end-of-treatment of a previous Phase 2 rusfertide study and are likely to continue benefiting from treatment with rusfertide based on their improved control of hematocrit levels <45% and reduced need for therapeutic phlebotomies. This study will provide long-term rusfertide treatment to these subjects and obtain data on safety and efficacy of long-term treatment with rusfertide.

ELIGIBILITY:
Inclusion Criteria:

* Subject who has completed at least 12 months of dosing with rusfertide and successfully completed the end of treatment visit of a previous Phase 2 study of rusfertide.
* Subject understands the study procedures, is willing and able to adhere to study requirements and agrees to participate in the study by giving written informed consent.

Key Exclusion Criteria:

* Subject who, in the opinion of the investigator, should not participate in the study.
* Subject who discontinue early from a previous rusfertide study for reasons other than enrolling in this study.
* Pregnant or lactating females.
* Women of childbearing potential (WOCBP) who do not agree to use medically acceptable contraception (<1% annual failure rate) during the study and for 30 days after the last dose of study drug.
* Men with partners of childbearing potential who do not agree to use medically acceptable contraception (<1% annual failure rate) during the study and for 90 days after the last dose of study drug.
* Men who do not agree to use a condom during the study and for 90 days after the last dose of study drug regardless of the partner's childbearing potential.
* A female subject intends to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 30 days after receiving the last dose of study drug.
* A male subject intends to donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after receiving the last dose of study drug.
* Plan to use investigational treatment other than rusfertide during the course of the study or within 28 days after last rusfertide dose.
* Subject with hypersensitivity to rusfertide or to any of the excipients.
* In the investigator's opinion the subject has progressive disease that cannot be managed by adjusting concurrent cytoreductive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Hematocrit | 0-2 years
  Median hematocrit
Phlebotomies | 0-2 years
  Number of phlebotomies

CONTACTS AND LOCATIONS:
Locations (1):
- Pontchartrain Cancer Care, Covington, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No